CLINICAL TRIAL: NCT05535309
Title: Epidemiological Study on Drug-induced Coagulation Disorder Caused by Cefoperazone Sulbactam Sodium and Construction of Prediction Model
Brief Title: Establishment of Risk Factors Model of Drug-induced Coagulation Disorder Caused by Cefoperazone Sulbactam Sodium
Status: Completed | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xiao Li，MD, Director, Qianfoshan Hospital
Other Study IDs: LCYY-LX-20220105
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-11

CONDITIONS: Risk Factors
Keywords: Coagulation disorder; Epidemiological study; Risk factors; Building models
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Occurrence of coagulation disorder: 1. All inpatients who used cefoperazone sulbactam sodium during hospitalization；
  2. Hospital stay ≥ 48h;
  3. Age ≥ 18 years old;
  4. Prothrombin time (PT), activated partial thromboplastin time (APTT), thrombin time (TT) and platelet (PLT) were detected twice or more during hospitalization
  Interventions: Drug: cefoperazone sulbactam sodium
- No coagulation disorder: 1. Inpatients who did not use cefoperazone sulbactam sodium during hospitalization;
  2. Hospital stay ≥ 48h;
  3. Age ≥ 18 years old;
  4. Prothrombin time (PT), activated partial thromboplastin time (APTT), thrombin time (TT) and platelet (PLT) were detected twice or more during hospitalization
  Interventions: Drug: cefoperazone sulbactam sodium

INTERVENTIONS:
Drug: cefoperazone sulbactam sodium — Cefoperazone sodium and Sulbactam Sodium for injection (1; 1) are white or almost white powder drugs, and the components are cefoperazone sodium and sulbactam sodium

SUMMARY:
The incidence rate of drug-induced blood diseases accounts for about 10% of all drug-induced diseases, most of which are serious at the time of onset, and the mortality rate can be as high as 32.5%. In this study, cefoperazone sulbactam sodium, which is commonly used in clinic, was selected as the target drug, and the epidemiological characteristics of drug-induced coagulation dysfunction and the construction of risk factor models were studied by single factor and multiple factor Logistic regression analysis.

DETAILED DESCRIPTION:
Investigators selected inpatients from Qianfoshan Hospital of Shandong Province from January 1, 2018 to December 30, 2021, extracted the cohort according to the inclusion and exclusion criteria, and divided it into exposure group and control group to find out the risk factors of cefoperazone sulbactam sodium causing coagulation disorders, and build a risk factor model of drug-induced coagulation disorders caused by cefoperazone sulbactam sodium.

ELIGIBILITY:
Inclusion Criteria:

All inpatients who used cefoperazone sulbactam sodium during hospitalization;

* Hospital stay ≥ 48h
* Age ≥ 18 years old

Exclusion Criteria:

* Age < 18 years
* Severe liver and kidney dysfunction
* Patients with vitamin K deficiency
* Patients with hematological diseases
* Patients with advanced malignant tumor or mental disease
* Patients with incomplete clinical data

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators included inpatients who were hospitalized from January 1, 2018 to December 30, 2021. The patients must be over 18 years old and take cefoperazone sulbactam sodium. Patients with underlying diseases that may affect the results were excluded and divided into exposure group and control group for study.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Coagulation disorder | Through study completion,up to half a year.
  Coagulation disorder occurred after cefoperazone sulbactam sodium was used in the patient's hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao Li,MD, Jinan, Shandong, China